CLINICAL TRIAL: NCT06766812
Title: Comparison of Dural Puncture Epidural Technique Versus Conventional Epidural Technique for Labour Analgesia in Primigravida;Comparative Randomized Double Blinded Study
Brief Title: Comparison of Dural Puncture Epidural Versus Conventional Epidural for Labour Analgesia in Primigravida
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Zidan, Resident-anesethiology department-sohag hospital university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh_Med__24_12_03Ms
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): dural puncture epidural technique in labour analgesia
  Interventions: Device: epidural set
- group B (Active Comparator): conventional epidural technique in labour analgesia
  Interventions: Device: epidural set

INTERVENTIONS:
Device: epidural set — The epidural space will be identified at either the L3-L4 or L4-L5 interspace using the loss of resistance technique with an 18 Gauge Epidural needle.A test dose of 3 mL of 2% lidocaine with epinephrine will be administered to each participant to rule out intravascular or intrathecal placement of the catheter. This ensures the proper placement of the catheter before the full dose of analgesia is administered.Following the test dose, an initial bolus of 8 mL of 0.25% bupivacaine combined with 2 μg/mL fentanyl will be administered to provide effective labor analgesia. Subsequently, maintenance Dose 0.125% 2 ml/0.5 hr

SUMMARY:
This study aims to compare the analgesic efficacy and safety of the Dural Puncture Epidural (DPE) technique versus the Conventional Epidural (CE) technique for labor analgesia in primigravida.

DETAILED DESCRIPTION:
The conventional epidural (CE) technique has been the gold standard for decades, providing continuous and adjustable pain relief during labor. However, the advent of new techniques, such as the Dural Puncture Epidural (DPE) technique, has led to ongoing research and debate over which method offers superior outcomes in terms of efficacy, onset of analgesia, maternal satisfaction, and safety.

The CE technique involves the placement of an epidural catheter into the epidural space, where local anesthetics and adjunctive drugs are administered to provide pain relief. While this technique is highly effective, it is not without limitations. Some parturients may experience a slow onset of analgesia, uneven drug distribution, or the need for frequent catheter adjustments, which can delay adequate pain relief and decrease maternal satisfaction . Furthermore, the CE technique has been associated with potential complications such as unilateral blocks, inadequate sacral analgesia, and the necessity for higher doses of local anesthetics, which may increase the risk of motor blockade and impact labor progression .

In contrast, the DPE technique is a novel approach that modifies the CE by incorporating an intentional dural puncture with a small-gauge spinal needle without administering intrathecal drugs. This modification is believed to facilitate the spread of epidurally administered drugs into the subarachnoid space, potentially enhancing the onset and quality of analgesia. The DPE technique aims to combine the benefits of both the CE and the Combined Spinal Epidural (CSE) techniques while minimizing their respective drawbacks, such as the hemodynamic instability associated with CSE and the slower onset of analgesia often seen with CE

ELIGIBILITY:
Inclusion Criteria:

1. Primigravida women aged 18-40 years.
2. Gestational age between 37 and 42 weeks.
3. Single pregnancy with vertex presentation.
4. Patients in active labor with cervical dilation of less than 5 cm at the time of epidural placement.
5. American Society of Anesthesiologist physical status I or II.
6. Patients who provide informed consent for participation in the study.

Exclusion Criteria:

1. Patients with contraindications to neuraxial anesthesia (e.g., coagulopathy, infection at the puncture site).
2. History of preeclampsia, gestational diabetes, or any other significant medical conditions that could influence labor or anesthesia outcomes.
3. Patients with a history of previous uterine surgery, including cesarean section.
4. Known fetal anomalies or non- vertex presentations.
5. Patients with morbid obesity (BMI > 40 kg/m²).
6. Allergy or hypersensitivity to local anesthetic-s used in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
onset of analgesia | 1 year
  be th
  e onset of effective Analgesia , defined
  as the time from the administration of the initial epidural bolus to a reduction in Visual Analogue Scale pain score to less than 3

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chau A, Bibbo C, Huang CC, Elterman KG, Cappiello EC, Robinson JN, Tsen LC. Dural Puncture Epidural Technique Improves Labor Analgesia Quality With Fewer Side Effects Compared With Epidural and Combined Spinal Epidural Techniques: A Randomized Clinical Trial. Anesth Analg. 2017 Feb;124(2):560-569. doi: 10.1213/ANE.0000000000001798. PMID 28067707
- [Background] Gunaydin B, Erel S. How neuraxial labor analgesia differs by approach: dural puncture epidural as a novel option. J Anesth. 2019 Feb;33(1):125-130. doi: 10.1007/s00540-018-2564-y. Epub 2018 Oct 6. PMID 30293143